CLINICAL TRIAL: NCT02839694
Title: Phase I Evaluation of Adjuvant Oral Decitabine and Tetrahydrouridine With or Without Celecoxib in Patients Undergoing Pulmonary Metastasectomy
Brief Title: Adjuvant Oral Decitabine and Tetrahydrouridine With or Without Celecoxib in People Undergoing Pulmonary Metastasectomy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160146; 16-C-0146
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-04-26

CONDITIONS: Neoplasm Metastasis; Sarcoma; Neoplasms, Germ Cell and Embryonal; Melanoma
Keywords: Lung Resection; Surgery; Bilateral Lung Metastases
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma; Neoplasms, Germ Cell and Embryonal; Melanoma | interventions — Decitabine; Tetrahydrouridine; Celecoxib

ARMS (3):
- Dose escalation cohort (Experimental): dose escalation cohort
  Interventions: Drug: decitabine (DAC); Drug: Tetrahydrouridine (THU)
- Expansion cohort (Experimental): expansion cohort at MTD
  Interventions: Drug: decitabine (DAC); Drug: Tetrahydrouridine (THU)
- expansion cohort with celecoxib (Active Comparator): expansion cohort at MTD with celecoxib
  Interventions: Drug: decitabine (DAC); Drug: Tetrahydrouridine (THU); Drug: Celecoxib

INTERVENTIONS:
Drug: decitabine (DAC) — Administered IV at increasing frequency or dose from 3-5 times per week for 8-12 weeks
Drug: Tetrahydrouridine (THU) — Administered IV at increasing frequency or dose from 3-5 times per week for 8-12 weeks
Drug: Celecoxib — 400 mg orally twice a day every day for while on DAC-THU therapy
  Arms: expansion cohort with celecoxib

SUMMARY:
Background:

Most patients who have surgery for cancer that has metastasized (spread) to the lungs later get more metastases that cannot be treated with surgery or chemotherapy. The drug resistance may be due to DNA changes in cancer cells that activate some genes and turn others off. Researchers want to test a combination of drugs for people with metasteses. Decitabine (DAC) may reverse the DNA changes. Tetrahydrouridine (THU) makes DAC last longer. Celecoxib may slow the progression of cancer.

Objectives:

To determine a safe dose of DAC and THU by mouth. To see if DAC-THU with or without celecoxib reactivates genes in lung metastases.

Eligibility:

Adults 18 years and older, with cancer in both lungs that can be treated with surgery.

Design:

Participants will be screened with:

Blood, lung, and heart tests

Scans

Tests for viruses

Pregnancy test

Participants will have blood and stool tests.

They will have surgery to remove metasteses in 1 lung.

About 3 weeks later, they will have lung scans. If the disease is not back, participants will get DAC and THU with or without celecoxib, by mouth for 6 weeks.

Participants will have more scans. If the disease is not worse, they will continue the study drugs for 4 more weeks.

Participants will have more scans and heart and lung tests. They will have surgery to remove metasteses from the other lung.

Participants will have weekly blood and urine tests, plus several blood draws the first 2 days of taking the drugs.

Participants will have exams and blood tests before each surgery.

Participants will have follow-up visits 1 and 3 months after the second surgery.

DETAILED DESCRIPTION:
Background:

* Whereas malignancies of diverse histologies express a variety of cancer testis antigens (CTAs), immune responses to these antigens appear uncommon in cancer patients, possibly due to low-level, heterogeneous antigen expression, as well as immunosuppressive regulatory T cells.
* In published studies we have demonstrated induction of NY-ESO-1 and MAGE-A3 in cancer cells of various histologies but not normal respiratory epithelial cells or fibroblasts following exposure to the DNA demethylating agent, Decitabine (DAC); up-regulation of these CTAs facilitated CTL-mediated lysis of tumor cells. We have also demonstrated eradication of pulmonary metastases in immunocompetent mice following systemic treatment with DAC and subsequent adoptive transfer of CTL recognizing the murine CTA, P1A. In a phase 1 trial, we demonstrated up-regulation of NY-ESO-1 and MAGE-A3 as well as reactivation of p16 in thoracic malignancies following intravenous 72hr DAC infusions. Chronic administration schedules are necessary for optimal gene induction in solid cancers.
* Additional studies using murine tumor models suggest that DNA demethylating agents may enhance the activity of immune checkpoint inhibitors not only by upregulating antigen presentation, but by inhibiting activity of myeloid derived suppressor cells (MDSC).
* Presently, there is no information regarding gene modulation and antitumor activity of oral epigenetic therapy in patients with solid tumors.
* In this study, the optimal frequency/dose of DAC-THU administration will be established in patients with bilateral pulmonary metastases, then an additional cohort of patients will receive DAC-THU together with celecoxib to inhibit activity of immunosuppressive Treg and myeloid derived suppressor cells. Correlative experiments will be performed to ascertain if oral epigenetic therapy modulates gene expression in pulmonary metastases and enhances antitumor immunity to these neoplasms.
* This trial is intended to establish the rationale and conditions for the use of oral DAC-THU +/- celecoxib in combination with immune checkpoint inhibitors or adoptive immunotherapy regimens targeting CTAs in patients with thoracic malignancies.

Objectives:

-To determine the pharmacokinetics, toxicities and maximum tolerated dose of oral DAC and THU with or without celecoxib in patients undergoing resection of pulmonary metastases

Eligibility:

* Patients with histologically or cytologically proven sarcoma, melanoma, germ cell tumors, or epithelial malignancies with bilateral pleuro-pulmonary metastases who can be rendered no clinical evidence of active disease (NED) or minimal residual disease (MRD) by metastasectomy.
* Patients greater than or equal to 18 years; ECOG performance status of 0-2, without evidence of unstable or decompensated myocardial disease; must have adequate pulmonary reserve evidenced by post-operative FEV1 and DLCO (Bullet) 40% predicted; pCO2 < 50 mm Hg and pO2 > 60 mm Hg on room air ABG; and be on no immunosuppressive medications except non-systemic corticosteroids.
* Patients must have a platelet count > 100,000, ANC greater than or equal to 1500 without transfusion or cytokine support, a normal PT, and adequate hepatic function as evidenced by a total bilirubin of < 1.5 times ULN. Serum creatinine less than or equal to 1.6 mg/ml or creatinine clearance > 70 ml/min/1.73m(2) at the time DAC/THU +/- celecoxib treatment commences.

Design:

* Eligible subjects with bilateral pulmonary metastases will undergo disease resection in one hemithorax
* Following recovery from initial hemithoracic metastasectomy (approximately 2-3 weeks), patients will begin oral DAC (0.2mg/kg)-THU (10 mg/kg) therapy 3-5 consecutive days/week depending on dose level. THU will be administered 60 minutes prior to DAC.
* If no dose limiting systemic toxicities (primarily myelosuppression) are observed, the frequency of DAC- THU will be sequentially increased to maximize intra-tumoral DNMT1 depletion while avoiding grade 3 or greater systemic toxicities.
* Once the frequency of DAC-THU therapy has been optimized, additional patients will also receive oral celecoxib (400mg PO BID).
* Oral DAC-THU +/- celecoxib therapy will continue for 6 weeks. Patients will then have repeat imaging studies. Those patients who exhibit no evidence of disease recurrence in the operated lung with disease progression in the contralateral hemithorax will undergo metastasectomy if there are no standard of care contraindications such as progression of disease in extrathoracic sites. Those patients exhibiting response to therapy evidenced by stable or regressing nodules will continue DAC-THU therapy for 4 additional weeks, followed by metastasectomy.
* Systemic toxicities and response to therapy will be recorded. Gene expression and DNA methylation profiles in pre- and post-treatment metastases will be compared to determine if DAC-THU therapy has altered the epigenome of the metastases. Serologic responses to upregulated CTAs as well as cell mediated responses to epigenetically-modified autologous EBV-transformed B and autologous tumor cells (if available) will be assessed before and after treatment if there is evidence of CT gene activation following DAC-THU +/- celecoxib treatment.
* DNMT and CTA expression levels in PBMC and tumor tissues will be evaluated before and after treatment to ascertain if DAC-THU depletes systemic DNMT levels, and to determine if alterations in DNMT/CTA expression in PBMC can serve as surrogates of respective drug induced changes in tumor tissues.
* Following complete metastasectomy, patients will be followed in the clinic with routine staging scans per standard of care guidelines.
* As the exact set of comparisons and analyses to be performed will be determined following completion of the trial, and will be based on limited numbers of patients, the analyses will be considered exploratory and hypothesis generating rather than definitive.
* Approximately 46 patients will be accrued to this trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with bilateral pulmonary metastases from sarcomas, melanomas, germ cell tumors, or epithelial malignancies metastatic to the lungs, mediastinum, or pleura who can be rendered no clinical evidence of active disease (NED) or minimal residual disease (MRD) by standard of care metastasectomy where NED refers to diagnostic tests failing to detect presence of disease and MRD refers to low-volume, subclinical disease which is not amenable to standard of care biopsy for histologic confirmation and poses no immediate threat to patient health and would not otherwise warrant standard of care treatment but surveillance instead.
* Patients must have a minimum of two metastases per hemithorax.
* Patients with active disease outside the thorax may be eligible for study once the extrathoracic disease is definitively treated by local modalities such as radiation, surgery, or radiofrequency ablation.
* Patients must have adequate pulmonary reserve evidenced by predicted post-operative FEV1 and DLCO equal to or greater than 40% predicted; pCO2 less than 50 mm Hg and pO2 greater than 60 mm Hg on room air ABG; and be on no immunosuppressive medications except inhaled corticosteroids.
* Patients must have received first line standard systemic therapy for their metastases (if applicable).
* Patients with intracranial metastases, which have been treated by surgery or radiation therapy, may be eligible for study provided there is no evidence of active disease and no requirement for anticonvulsant therapy or steroids following treatment.
* Patients must have an ECOG performance status of 0-2.
* Patients must have recovered from non-hematologic toxicities associated with treatment of malignancy to less than or equal to grade 1.
* Patients must be 18 years of age or older due to the unknown effects of systemic DNA hypomethylation and immunologic responses to germ cell-restricted gene products during childhood and adolescent development.
* Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

  * Absolute neutrophil count greater than 1500/mm(3) without transfusion or cytokine support
  * Platelet count greater than 100,000/mm(3)
  * Hemoglobin greater than 8g/dl (patients may receive transfusions to meet this parameter)
  * PT no more than 2 seconds above the ULN
  * Total bilirubin <1.5 times upper limits of normal
  * Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2).
* Seronegative for HIV antibody. Note: The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment.
* Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Patients must be aware of the neoplastic nature of their illnesses, the experimental nature of the therapy, alternative treatments, potential benefits, and risks.
* Patients must be willing to practice birth control during and for four months following treatment.
* Patients must be able to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening or otherwise altering the product formulation.
* Patients who had prior lung resection are eligible provided they fulfil the rest of the eligibility criteria.
* Patients must be willing to sign an informed consent.

EXCLUSION CRITERIA:

* Patients with uncontrollable progression of extra-thoracic disease will be excluded from study.
* Patients requiring corticosteroids (other than inhaled) will be excluded.
* Patients receiving warfarin anticoagulation, who cannot be transferred to other agents such as enoxaparin or dabigatran, and for whom anticoagulants cannot be held for up to 24 hours will be excluded.
* Patients with uncontrolled hypertension (>160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated CHF (>NYHA Class II), or myocardial infarction within 6 months of study will be excluded.
* Patients with other cardiac diseases may be excluded at the discretion of the PI following consultation with Cardiology consultants.
* Pregnant and/or lactating women will be excluded due to the unknown, potentially harmful effects of immune response to CT-X antigens and stem cell proteins that may be expressed in placenta, fetus, and neonates.
* Patients with active infections, including HIV, will be excluded, due to unknown effects DAC/THU on systemic immunity.
* For patients enrolled on celecoxib cohort: history of ulcer disease or gastrointestinal bleeding, hypersensitivity or asthma to celecoxib, sulfa drugs, aspirin or other NSAID.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-07; Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 weeks after the start of study therapy
Table of toxicities including type, severity, time of onset, time of resolution and probable association with study regimen | 30 days after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)